CLINICAL TRIAL: NCT05796778
Title: Sub Omohyoid Suprascapular Nerve Block Versus Interscalene Nerve Block for Postoperative Shoulder Surgery Pain: Randomized Comparative Study.
Brief Title: Sub Omohyoid Suprascapular Nerve Block Versus Interscalene Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 685/2023
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pain; Regional Anesthesia; Nerve Block
Keywords: Interscalene brachial plexus block; shoulder pain; subomohyoid plane block
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subomohyoid suprascapular nerve (Experimental): superficial probe of ultrasound was placed in the transverse plane to visualize the superior trunk in the short axis. The suprascapular nerve was identified as it branched off from the superior trunk and traced until it coursed beneath the inferior belly of the omohyoid muscle.
  Interventions: Procedure: subomohyoid plane block
- Interscalene brachial plexus (Active Comparator): ultrasound-guided interscalene block involves imaging the C5 and C6 roots at approximately the level of the cricoid cartilage, just distal to where they emerge from behind their respective transverse processes and where they lie in the groove between the anterior and middle scalene muscles
  Interventions: Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Procedure: subomohyoid plane block — The block needle was inserted in line with the probe in a lateral-to-medial orientation toward the suprascapular nerve. Local anesthetic solution was then injected after negative aspiration for blood to achieve circumferential spread around the neurovascular bundle
  Arms: subomohyoid suprascapular nerve
Procedure: Interscalene brachial plexus block — The block needle is usually advanced in plane in a lateral-to-medial direction through the middle scalene muscle to contact the nerve roots and inject local anesthetic around them.
  Arms: Interscalene brachial plexus

SUMMARY:
Shoulder surgery can be very painful surgery after which the use of opioids is often required. The well-known side-effects of opioids (e.g. respiratory depression, somnolence, nausea, vomiting, and pruritus) limit their use in so called 'fast track' surgery and anaesthesia programmes.

the study aimed to compare the effect of sub omohyoid suprascapular nerve block versus interscalene nerve block in preventing postoperative pain and decreasing analgesic consumption in patients scheduled for shoulder surgery

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years.
2. ASA I-II.
3. Both sexes.
4. Shoulder surgery.

Exclusion Criteria:

1. Patient refusal
2. Allergy to local anesthetics
3. BMI >40 kg/m2
4. Bleeding diathesis or history of anticoagulant use.
5. Psychiatric diseases.
6. Infection of the skin at the site of needle punctures area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain score | 24 hour
  pain score from 0 to 10 which mean 0 no pain and 10 the worst pain ever

SECONDARY OUTCOMES:
Time of first analgesic request | 24 hour
  the time of first demand rescue analgesia
Total analgesic consumption | 24 hour
  total fentanyl demand
Incidence of any side effects | 24 hour
  oxygen desaturation, pneumothorax, dyspnea, and phrenic nerve palsy, block, and opioid-related side effects

CONTACTS AND LOCATIONS:
Overall Officials: hassan m. hetta, lecturer, Principal Investigator — Minia University, faculty of medicine
Locations (1):
- Minia University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No